CLINICAL TRIAL: NCT07363629
Title: Impact of Preserving Versus Ligating the Right Gastric Artery on Anastomotic Outcomes After McKeown Esophagectomy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yongbin Song, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20200507
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RGA Preservation Group (Experimental): Patients in this arm underwent McKeown MIE where the stomach was mobilized while carefully preserving the main trunk of the right gastric artery (RGA). Lymph nodes along the lesser curvature (Station 3) were dissected by peeling them away from the vascular arcade.
  Interventions: Procedure: McKeown MIE with RGA Preservation
- RGA Ligation Group (Active Comparator): Patients in this arm underwent McKeown MIE where the right gastric artery (RGA) was identified at its origin from the proper hepatic artery and ligated at the root to facilitate en bloc resection of Station 3 lymph nodes.
  Interventions: Procedure: McKeown MIE with RGA Ligation

INTERVENTIONS:
Procedure: McKeown MIE with RGA Preservation — Patients in this arm underwent McKeown MIE where the stomach was mobilized while carefully preserving the main trunk of the right gastric artery (RGA). Lymph nodes along the lesser curvature (Station 3) were dissected by peeling them away from the vascular arcade.
  Arms: RGA Preservation Group
Procedure: McKeown MIE with RGA Ligation — Patients in this arm underwent McKeown MIE where the right gastric artery (RGA) was identified at its origin from the proper hepatic artery and ligated at the root to facilitate en bloc resection of Station 3 lymph nodes.
  Arms: RGA Ligation Group

SUMMARY:
This randomized controlled trial evaluates the impact of preserving versus ligating the Right Gastric Artery (RGA) on postoperative anastomotic complications in patients undergoing McKeown minimally invasive esophagectomy (MIE) for esophageal squamous cell carcinoma. Specifically, the study compares the incidence of anastomotic leakage and stenosis between two groups of patients reconstructed with a 3cm-wide gastric conduit.

DETAILED DESCRIPTION:
Anastomotic leakage (AL) and benign anastomotic stenosis (BAS) are critical complications following McKeown MIE. While the right gastroepiploic artery (RGEA) is the primary blood supply for the gastric conduit, the role of the Right Gastric Artery (RGA) remains controversial. Some evidence suggests preserving the RGA may improve perfusion to the proximal gastric conduit, potentially reducing ischemic complications. In this single-center prospective RCT, 120 eligible patients were randomized 1:1 into an RGA Preservation Group (Group A) and an RGA Ligation Group (Group B). Both groups underwent reconstruction with a narrow (3cm) gastric conduit. The study aims to provide evidence on whether RGA preservation improves hemodynamic outcomes as manifested by reduced leakage and stenosis rates.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the middle or upper thoracic esophagus.
* Candidates for elective McKeown minimally invasive esophagectomy (MIE).
* Age 18-75 years.
* Preoperative clinical stage I-IIIA (cT1-3N0-1M0) according to the AJCC/UICC 8th Edition TNM staging system.

Exclusion Criteria:

* Clinical stage IIIB or IV.
* History of previous thoracic or abdominal surgery affecting the stomach or esophagus.
* Neoadjuvant chemoradiotherapy (to eliminate confounding effects on tissue healing).
* Severe comorbidities (e.g., uncontrolled diabetes, severe cardiopulmonary dysfunction, liver cirrhosis).
* Intraoperative finding of unresectable tumor.
* Conversion to open surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Cervical Anastomotic Leakage | Up to 30 days postoperatively
  Defined as the extravasation of contrast on esophagogram or the presence of saliva/gastric content in the cervical wound, often accompanied by fever or inflammatory signs.
Incidence of Anastomotic Stenosis (Early) | 2 months postoperatively
  Assessment of benign anastomotic stenosis (BAS) via gastroscopy and contrast swallow. Stenosis was graded based on luminal diameter and dysphagia symptoms.
Incidence of Anastomotic Stenosis (Late) | 4 months postoperatively
  Assessment of benign anastomotic stenosis (BAS) via gastroscopy and contrast swallow. Stenosis was graded based on luminal diameter and dysphagia symptoms.

SECONDARY OUTCOMES:
Operative Time | Day 1 (Day of Surgery)
  The total duration of the surgical procedure measured in minutes.
Lymph Node Yield | Day 1 (Day of Surgery)
  The total count of lymph nodes harvested during the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei General Hospital, Shijiazhuang, Hebei, China